CLINICAL TRIAL: NCT06685562
Title: The 4D PICTURE Project - Design-based Data-driven Decision-support Tools: Producing Improved Cancer Outcomes Through User-Centered Research
Brief Title: The 4D PICTURE Project: Evaluating Metro Mapping As a Method to Support Shared Decision Making in Oncology
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Sint Franciscus Gasthuis (Other); Vejle Hospital (Other); Hospital Miguel Servet (Other); Medical Center Haaglanden (Other)
Responsible Party: Principal Investigator, amstiggelbout, Prof. Dr. Anne M. Stiggelbout, Leiden University Medical Center
Other Study IDs: 8423
Record Dates: First submitted 2024-10-31; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Patients; Melanoma Cancer; Prostate Cancer; Supportive Care in Cancer
Keywords: MetroMapping; Shared Decision Making; Oncology; Service design; care path redesign
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-test patients: Prostate cancer patients, breast cancer patients, and melanoma patients from Spain, Denmark and the Netherlands recruited in the pre-test phase to observe care as usual
- Post-test patients: Prostate cancer patients, breast cancer patients, and melanoma patients from Spain, Denmark and the Netherlands recruited in the pre-test phase to observe care with the implementation of MetroMapping

SUMMARY:
The goal of this observational study is to evaluate the impact of MetroMapping (a service design methodology) on Shared Decision Making in cancer care paths. The goal is to improve Shared Decision Making and make cancer care paths less overwhelming. The study will include adult participants (older than 18 years) with breast, prostate and melanoma cancers. The main question is How does the implementation of MetroMapping improve Shared Decision Making in cancer care paths.

500 patients, across the Netherlands, Spain, and Denmark, will be enrolled in a pre- and posttest phase. Including 100 breast cancer, 100 prostate cancer, and 50 melanoma patients per phase. To further understand patient experiences, the researchers will audio-record and transcribe the Shared Decision Making consultation of a subset of participants (10 per tumor type per country). A total of 120 audio-recordings across both study phases will be collected. In the post-test phase, a personal care path navigator will be created and the researchers will conduct interviews with 3 patients per care path and interviews with clinicians (12 per country, a total of 36) to assess their experiences with MetroMapping.

The study is a pre-test and post-test multiple methods design, gathering both quantitative and qualitative data across care paths in the Netherlands, Spain and Denmark. Quantitative data will be collected via electronic (Castor EDC & RedCap) and paper questionnaires. Participants will receive the first set of questionnaires, one week after their decision-making consult. Encompassing the following questionnaires (I-SHARE for perceived Shared Decision Making, Control Preferences Scale for the perceived roles in the actual decision, Decisions Made, Decisional Comfort Scale, SCIP B Information Provision, PEPPI-5 Perceived Efficacy in Patient-Physician Interactions, Trust in Oncologists, Health Literacy) and for the cost-effectiveness analysis for our partner (UMIT TIROL) the EORTC QLU C10-D and EQ-5D5l will be added to assess utilities. In the post-test participants will receive the second set of questionnaires, 6 months after the first set of questionnaires. This set encompasses (Healthcare Integration INTEGrate, Person Centered Coordinated Care Experiences P3CEQ, Decisional Regret Scale, Trust in Oncologists, EORTC QLU-C10D, EQ-5D5L, Productivity Cost Questionnaires.

This study includes a pre-implementation comparison group, and results will be compared with post-implementation outcomes.

Participants will complete the questionnaires and provide demographic and clinical data (consent for sharing medical file is asked) and an audio-recording of their consultation will be made. Participants in the post-phase will participate in interviews about their experiences with the implementation of MetroMapping.

The audio-recordings will be transcribed and analyzed using the OPTION and 4SDM coding instruments. Data will be analyzed using both univariate and multivariate statistical methods. Transcript of audio-recordings will be analyzed using thematic analysis and the coding instruments.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) (either being the patient or the informal caregiver in the care path)
* Prostate cancer, breast cancer or melanoma cancer
* Able to provide consent
* Able to speak Dutch, Danish, Spanish, Catalan

Exclusion Criteria:

A potential subject who does not meet any of the above criteria will be excluded from participation in this study. There are no further specified exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult participants aged 18 years and older. The participants will be recruited from specific hospital in three countries:
  Prostate cancer patients: Sint Franciscus Gasthuis in Rotterdam, the Netherlands & Lillebaelt Hospital in Vejle, Denmark Melanoma patients: Leiden University Medical Center in Leiden, the Netherlands, Haaglanden Medical Center in The Hague, the Netherlands & Miguel Servet University Hospital in Zaragoza, Spain.
  Breast cancer patients: Lillebaelt Hospital in Vejle, Denmark & Miguel Servet University Hospital in Zaragoza, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
The impact of MetroMapping on perceived Shared Decision Making | The time frame is one week after the decision making consultation
  To test the impact of MetroMapping on perceived Shared Decision Making. The iSHARE questionnaire for perceived shared-decision making will be used. The questionnaire assesses Shared Decision Making in oncology. The iSHARE has 15 items with dimension scores (0-5) and a total score (0-30). Higher dimension and total scores indicate higher levels of Shared Decision Making.

SECONDARY OUTCOMES:
The impact of MetroMapping on the decision-making process | Patients will receive the questionnaires one week after their consultation and 6 months after the consultation.
  To evaluate the effect of MetroMapping on the decision-making process various outcomes will be used.
  * The Control Preferences Scale (CPS) for the perceived roles in actual decision. The CPS is a single-item 5 point scale (0-4) ranging from passive to active.
  * Decisions Made, an open-ended question to gain insight into the final treatment choice.
  * Decisional Conflict Scale (DCS) is a 16 item questionnaire on a 5 point scale. Total score range from 0 [feels extremely certain about best choice] to 100 [feels extremely uncertain about best choice].
  Decisional Regret Scale is a 5 item questionnaire on a 5 point scale, ranging from 1 (strongly agree) to 5 (strongly disagree). A higher number will indicate more regret.

OTHER OUTCOMES:
The evaluation of MetroMapping on the care path | Patients will receive the questionnaires one week after their consultation and 6 months after the consultation.
  To evaluate the impact of MetroMapping on the carepath several outcomes will be tested. Satisfaction with Cancer Information Profile (SCIPB) is an 7 item questionnaire on a 5 point scale (5-1). Total score ranges from 7-35. Higher score indicating a higher satisfaction with information. Perceived efficacy in Patient-Physician Interactions is a 5 item questionnaire on a scale of 1 to 5. Range of possible scores is (5-25). 25 meaning the highest patient self-efficacy. Trust in Oncologists is an 18 item questionnaire on a 5-point scale (1 to 5). Scores ranging from 18 to 90. A higher score indicates a higher level of trust in the oncologist. Health Literacy is an 3 item questionnaire. Scores ranging from 1 to 5. A higher score indicates a higher level of health literacy. Healthcare Integration (integRATE) is an 4 item questionnaire (0-3) with higher values indicating more integration Person Centered Coordinated Care Experiences (P3CEQ) is an 11 item questionnaire.

CONTACTS AND LOCATIONS:
Locations (3):
- Sygehus Lillebaelt, Vejle, Denmark
- Leiden University Medical Center, Leiden, Netherlands
- Miguel Servet University Hospital, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No